CLINICAL TRIAL: NCT04342429
Title: RAD4649-19: Prospective Study of Intensity-Modulated Proton Therapy (IMPT) for Small Cell Lung Cancer
Brief Title: Prospective Study of Intensity-Modulated Proton Therapy (IMPT) for Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sibo Tian, Principal Investigator, Associate Professor, Department of Radiation Oncology, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00110109
Record Dates: First submitted 2020-03-24; First posted 2020-04-13 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prospective Study of Intensity-Modulated Proton Therapy (IMPT) (Experimental): This is the first prospective study to investigate the safety and efficacy of IMPT for the treatment of SCLC. We will utilize adaptive planning throughout the radiation course. In addition, we will study the dosimetric parameters of IMPT and their correlation with treatment-related toxicities, particularly cardiac events.
  Interventions: Radiation: Proton-beam Therapy for Small Cell Lung Cancer

INTERVENTIONS:
Radiation: Proton-beam Therapy for Small Cell Lung Cancer — The goal of intensity-modulated proton therapy (IMPT) is to deliver radiation to the tumor while minimizing exposure to surrounding normal tissues.

SUMMARY:
To assess the safety and efficacy of intensity-modulated proton therapy (IMPT) for small cell lung cancer (SCLC)

DETAILED DESCRIPTION:
To determine the optimal schedule for three-dimensional verification imaging and necessary re-planning of patients undergoing IMPT for a rapidly changing tumor (small cell lung cancer).

* To determine the rate of cardiac toxicities from IMPT in patients with small cell lung cancer compared with historical controls receiving photon-based treatment.
* To determine the rate of pneumonitis and esophagitis from IMPT and compare with historical controls receiving photon based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed small cell lung cancer, limited or extensive stage.
* Patients who are offered thoracic radiotherapy with intensity-modulated proton therapy (IMPT) techniques delivering 30-66 Gy in 15-33 fractions at 2 Gy per fraction, at the recommendation of the treating radiation oncologist.
* Age 18 or greater

Exclusion Criteria:

* Prior radiation therapy which would provide significant dose overlap with the planned target volume(s)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Patients with small cell lung cancer (SCLC) will be assessed with the intensity-modulated proton therapy (IMPT). | Up to 1 year from study start
  Patients enrolled will experience <35% incidence of cardiac events at 1-year. Cardiac events included are acute heart disease, acute myocardial infarction, cardiomyopathy, dysrhythmia, heart failure, pericarditis, and pericardial effusion.
Determination of the optimal frequency of conebeam CT during treatment and subsequent need for adaptive re-planning | Up to 1,2, and 5 years
  The optimal frequency of conebeam CT during treatment will be determined by a mixed model:
  * The local control, distant metastases, patterns of failure will be summarized as frequency and percentage.
  * Chi-square test will be used to test their relationships with other categorical variables.
  * General linear model will be used to measure their association with continuous covariates with and without adjusting for other factors

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Higgins, MD, Principal Investigator — Emory University-Winship Cancer Institute
Locations (1):
- Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04342429/Prot_SAP_000.pdf